CLINICAL TRIAL: NCT02043210
Title: Computer Based Training in CBT for Spanish-speaking Substance Users
Brief Title: CBT for Spanish Speakers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1110009151; 1R01DA030369-01A1 (NIH)
Record Dates: First submitted 2014-01-10; First posted 2014-01-23 (Estimated); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Substance Use
Keywords: substance use, Spanish speaking, CBT4CBT
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Treatment as Usual (Active Comparator): Treatment that would normally be received at the clinic typically consisting of individual or group counseling sessions focusing on substance abuse.
  Interventions: Behavioral: Standard Treatment as Usual
- CBT4CBT plus Standard treatment as usual (Experimental): A computerized program that teaches skills for stopping substance use by increasing coping skills such as how to understand patterns of drug use, coping with cravings, etc. plus standard treatment as usual.
  Interventions: Behavioral: CBT4CBT plus Standard treatment as usual

INTERVENTIONS:
Behavioral: Standard Treatment as Usual — Treatment normally offered at this clinic which could include individual or group substance use counseling sessions one time per week lasting one hour each time.
  Arms: Standard Treatment as Usual
Behavioral: CBT4CBT plus Standard treatment as usual — Subjects work with a computerized program in Spanish that teaches skills for stopping substance use and increasing coping skills. Computerized sessions are one time per week and last about one hour per session. Plus Standard treatment as usual
  Arms: CBT4CBT plus Standard treatment as usual

SUMMARY:
The investigators are conducting a randomized clinical trial of our new web-based version of the CBT4CBT (Computer Based Training for Cognitive Behavioral Therapy) in Spanish. This program specifically designed for Spanish-speaking substance users to evaluate its effectiveness relative to standard outpatient counseling at the Hispanic Clinic. The computer-based training program (CBT4CBT) focuses on teaching basic coping skills, presenting examples of effective use of coping skills in a number of realistic situations in video form, and providing opportunities for patients to practice and review new skills while receiving substance use treatment.

DETAILED DESCRIPTION:
100 Spanish-speaking substance using individuals seeking treatment at the Hispanic Clinic of the Connecticut Mental Health Center will be randomized to (1) standard outpatient counseling at the Hispanic Clinic (typically consisting of weekly group counseling), OR (2) CBT4CBT plus standard outpatient counseling. Treatments will be delivered over an 8-week period with a six-month follow-up after termination of the study treatments. The primary outcome measures will be reduction in substance use (frequency of substance use by time, confirmed by urine toxicology screens and breathalyzers). Secondary outcomes will include treatment utilization and cost, several measures intended to detect whether web-based CBT4CBT retains key characteristics of traditional clinician-administered CBT (e.g., acquisition of coping skills, use of change strategies), participant characteristics which will be evaluated as potential moderators of outcome, as well as participant satisfaction and treatment credibility.

ELIGIBILITY:
Inclusion Criteria:

* Are 18 years of age or older.
* Are applying for outpatient, non-agonist substance abuse treatment at the Hispanic Clinic.
* Meet current DSM-IV criteria for cocaine, marijuana, opioid, alcohol or other stimulant abuse or dependence.
* Are sufficiently stable for 8 weeks of outpatient treatment.
* Can commit to 8 weeks of treatment and are willing to be randomized to treatment
* Are willing to provide locator information for follow-up.
* Speak Spanish as their preferred or principal (most commonly spoken)language

Exclusion Criteria:

* Have an untreated bipolar or schizophrenic disorder.
* Who have a current legal case pending such that incarceration during 8-week protocol is likely.
* Are physically dependent on alcohol, opioids or benzodiazepines

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2014-01; Primary Completion 2017-08 (Actual); Study Completion 2017-09-11 (Actual)

PRIMARY OUTCOMES:
Reduction in substance use | 8 weeks
  Reduction in substance use will be measured by Time Line Follow back self report and urine toxicology screening

SECONDARY OUTCOMES:
Subjects ability to demonstrate coping skills through a computerized role-playing evaluation and homework | 8 weeks
  Computerized role-playing will be used to demonstrate ability to use learned coping skills in various settings.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Carroll, PhD, Principal Investigator — Yale University
Locations (4):
- United States (4):
  - Fair Haven Community Health, New Haven, Connecticut
  - MAAS, New Haven, Connecticut
  - Hispanic Clinic, New Haven, Connecticut
  - Substance Abuse Treatment Unit (SATU), New Haven, Connecticut

REFERENCES:
- [Derived] Benitez B, Frankforter T, Nich C, Paris M, Kiluk BD. Comparing content within a culturally-adapted digital treatment for Hispanic patients with alcohol use disorder. NPJ Digit Med. 2025 Dec 8;9(1):23. doi: 10.1038/s41746-025-02197-7. PMID 41361015